CLINICAL TRIAL: NCT02723799
Title: Promoting Hope at the End of Life: Effectiveness of a Hope Intervention Program in Palliative Patients
Brief Title: Hope Promotion Program: Effectiveness in Palliative Patients
Acronym: HPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Leiria (Other)
Collaborators: Universidade Católica Portuguesa (Other)
Responsible Party: Principal Investigator, Ana Querido, PhD, Instituto Politécnico de Leiria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ana Querido - IPLeiria
Record Dates: First submitted 2016-03-14; First posted 2016-03-30 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Chronically Ill
Keywords: Hope; Quality of Life; Comfort
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hope Promotion Program (HPP) (Experimental): Plus to the standard treatment protocol, all the participants in this group attend the HPP, consisting of a three individual session's carried out by the nurse in patients' homes. It includes viewing the film Hopeful Living, enrolling in a hope activity from the Hope activity book, a relaxation activity and a negotiated plan to exercise hope in a regular basis.
  Interventions: Behavioral: Hope Promotion Program (HPP); Other: Standard Treatment Protocol
- Standard Treatment Protocol (Other): Participants in this group has not access to a hope intervention. Data collection for outcome variables is the same as the participants in the other arms.
  Interventions: Other: Standard Treatment Protocol

INTERVENTIONS:
Behavioral: Hope Promotion Program (HPP) — HPP is based on literature review and qualitative research in hope at the end-of-life. The film "Hopeful living" reflects the findings of the grounded theory study. Hope activity book is the final product of the literature review on hope interventions and its activities were tested in their feasibility and suitability in our previous research with persons with advanced cancer and their families.
  Arms: Hope Promotion Program (HPP)
Other: Standard Treatment Protocol — Regular assessment and care by the hospital outpatient health care team.

SUMMARY:
This study aims to:

I. Develop and pilot test the effectiveness of a Hope Promotion Program compared with the standard treatment protocol, in hope, comfort and quality of life, based on a population of palliative patients followed at Oncology day care unit.

II. Evaluate perceptions and acceptability of Hope Promotion Program among palliative patients submitted to the intervention program.

DETAILED DESCRIPTION:
Background: Hope is essential in the experience of living with advanced chronic disease. Maintaining hope in situations of physical, psychological, spiritual and social suffering requires expertise and can be very difficult to achieve without the help of professionals, leading to hopelessness, despair and desire to hasten death (Rodin et al., 2007;Breitbart, 2000; Monforte-Royo, et al., 2012) The research team has designed an intervention program - Hope Promotion Program (HPP) to increase hope, comfort and quality of life in palliative patients. HPP consists of a three session's individual interventions carried out by the researcher in patients homes. The first session includes viewing the film Hopeful Living, produced by the research team, inspired by Duggleby et al, (2007) which features palliative patients, caregivers and health professionals describing their experiences of hope. The second session consists of patients' expression of feelings and emotions related with experience of living with a chronic advanced disease and the choice of a hope activity from the Hope activity book - a collection of hope activities specially designed for people living with an advanced chronic disease. The third session includes a relaxation activity and a plan to include hope exercise in patients' activities of daily living.

This project was designed according to the literature review of hope interventions and have the potential to become part of palliative care interventions evidenced based.

Aims: The purpose of this study is to evaluate the acceptability and feasibility and collect preliminary data on the effectiveness of the Hope Promotion Program for persons in palliative situation residing at home.

Moreover this project will allow to a) Obtain relevant information about hope, comfort and quality of life of palliative patients; b) Tailor therapeutic strategies to individual needs; c) increase hope, comfort and quality of life in patients at the end of life.

Sample: Patients with a chronic advanced disease in palliative situation, recruited from Oncology day care units of two district hospital in the centre of Portugal. Inclusion criterion for participants are: a) 18 years of age and older, b) Portuguese speaking, c) have cognitive capacity to participate in the study (MMSE>15) and d) have agreed to participate in the study. An interview with a nurse precede the inclusion in the study to explain the study and obtain written informed consent.

Design: This study is designed as a mix-methods randomized clinical trial (Quantitative +Qualitative) design. Patients eligible, are randomly assigned to one of two groups: 1) treatment (Hope Promotion Program delivered by a nurse in three sessions during one week), 2) usual care group.

In all groups, demographic information and measures of hope (Herth Hope Index), quality of life (McGillQOL), Comfort (Hospice Comfort Questionnaire) will be collected by a trained research nurse at baseline, day 15 and one month. Participants in group 1 (treatment group) will be asked to describe what they were thinking about when doing the hope activities on day 15 and one month using qualitative interviews. At one month all participants will be interviewed using open ended audiotaped questions to help evaluate the program and study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Portuguese speaking
* Have a chronic advanced disease non-responding to treatment, metastatic disease, episodes of non-controlled symptoms
* Have health care assistance by a health care team in an outpatient setting
* Cognitive ability to answer the questionnaires (MMSE>15 for illiterate participants, >22 for participants with 11 years of schooling, >27 for participants with more than 11 years of schooling)
* Consenting to voluntarily participate in the study.

Exclusion Criteria:

* Patients with high suffering from uncontrolled and recurrent presence of symptoms (nausea, vomiting, pain),
* Patients with performance status under 30, due to their particularly vulnerability, intervention would need energy required to vital functions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Hope measured by the Portuguese version of Herth Hope Index | Change from baseline at day 15 and 30
  Hope is measured by the Portuguese version of Herth Hope Index for chronic conditions (HHI-PT-DC). The HHI-PT-DC is a 10 item (1-4 point) Likert scale that delineates two sub-scales of hope: a) temporality, trust and interconnection, b) positive readiness and expectancy. The HHI-PT-DC takes approximately 5 minutes to complete. Summative scores range from 10-40, with a higher score denoting greater hope.

SECONDARY OUTCOMES:
Comfort measured by Portuguese version of Hospice Comfort Questionnaire | Change from baseline at day 15 and 30
  Comfort is measured by Portuguese version of Hospice Comfort Questionnaire, based on holistic comfort questionnaire, developed by Kolcaba (HCQ-PT-DC). This instrument is composed by 26 items (1-6 points) Likert-scale that addresses the three states of comfort: relief, ease and transcendence. The higher the score, the higher the subjects' reported comfort.
Quality of Life measured by the Portuguese version of McGill Quality of Life Questionnaire (MQOL-PT-DC) | Change from baseline at day 15 and 30
  Quality of Life is measured by the Portuguese version of McGill Quality of Life Questionnaire (MQOL-PT-DC). The MQOL-PT-DC is a quality of life assessment measure reflecting 4 domains of quality of life: physical health, psychological symptoms, existential well-being, and support. The MQOL-PT-DC is comprised of 16 items, assessed in a self-rating numerical scale (0-10) and Single Item Scale (0-10) to assess subjective quality of life. Higher scores indicates better QOL.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryan RE, Connolly M, Bradford NK, Henderson S, Herbert A, Schonfeld L, Young J, Bothroyd JI, Henderson A. Interventions for interpersonal communication about end of life care between health practitioners and affected people. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD013116. doi: 10.1002/14651858.CD013116.pub2. PMID 35802350